CLINICAL TRIAL: NCT05601245
Title: High Voltage Pulsed Current Versus Microcurrent Stimulation Therapy in the Treatment of Chronic Wounds
Brief Title: High Voltage Pulsed Current and Microcurrent Stimulation Therapy in Treatment of Wounds.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Shaimaa Mohamed Ahmed Elsayeh, Lecturer of physical therapy, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/003742
Record Dates: First submitted 2022-10-08; First posted 2022-11-01 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Wound; Ulcer
Keywords: High-voltage pulsed current; Micro-current therapy; Chronic wound
MeSH Terms: conditions — Wounds and Injuries; Ulcer

STUDY DESIGN:
Intervention Model Description: Sixty patients (male and female) with chronic wounds (pressure ulcers) does not heal within six weeks were involved in the study.
  The diagnosis will be made clinically by the physician. The patients will be randomly assigned into two equal groups in number, two study groups (one for high-voltage pulsed galvanic current and the other for microcurrent therapy). Both groups will receive the same traditional physical therapy routine and conservative treatment for the wound for six weeks.
Who Masked: Outcomes Assessor
Masking Description: Closed envelop method
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High voltage pulsed current (Experimental): Twenty patients with chronic wounds will be managed by the high-voltage pulsed current for 45 as the total treatment duration and the polarity will be reversed after 22 minutes, three sessions per week for six weeks.
  Interventions: Other: High voltage pulsed current
- Microcurrent therapy (Experimental): Twenty patients with chronic wounds will be managed by microcurrent therapy for 40 minutes, three sessions per week for six weeks.
  Interventions: Other: Microcurrent therapy

INTERVENTIONS:
Other: High voltage pulsed current — The treatment session duration is 45 minutes (Reverse the polarity after the first 22 minutes)
  Other Names: Conventional physical therapy program
  Arms: High voltage pulsed current
Other: Microcurrent therapy — The treatment session duration is 40 minutes.
  Other Names: Conventional physical therapy program
  Arms: Microcurrent therapy

SUMMARY:
The purpose of this study is to evaluate the effectiveness of high-voltage pulsed current (HVPC) and microcurrent stimulation therapy (MST) in treating chronic wounds and to compare their effects.

DETAILED DESCRIPTION:
Sixty patients with chronic wounds (pressure ulcers) and their ages will be ranged from 45 to 60 years old. They will be recruited from the outpatient clinic at Kasr Al-Aini Hospitals and they will be randomly assigned into two groups of equal numbers, each one will contain thirty patients. High-voltage pulsed current group and microcurrent stimulation therapy groups. The change in wound surface area and wound volume will be measured before the intervention and after six weeks of intervention.

ELIGIBILITY:
Inclusion Criteria:

* Patients are of both sexes.
* Subject's age will be from 45 to 60 years.
* All patients will enter the study having their informed consent.
* All patients will be assessed by a physician before starting the study procedure.
* All patients suffer from a chronic wound not healed more than or within six weeks.

Exclusion Criteria:

* Patients with acute wounds.
* Patients with burn wound injuries.
* Malignancy in the wound.
* Necrotic tissue in the wound.

Ages: 45 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2022-08-10 (Actual); Primary Completion 2023-04-28 (Actual); Study Completion 2023-07-20 (Actual)

PRIMARY OUTCOMES:
Change in wound surface area | Baseline and six weeks after the intervention.
  A sterilized transparency film will be placed over the ulcer. The ulcer perimeter was traced by using the film tipped transparency marker. Each ulcer was traced three times to establish measurement reliability. After tracing, the side of the transparency film facing the ulcer will be cleaned with a piece of cotton and alcohol. Carbon paper was placed over the 1-mm-squared metric graph paper. The traced transparency film was placed over the carbon paper with white paper in between and the tracing will be transcribed onto the metric graph paper. WSA was calculated by counting the number of square millimeters on the metric graph within the wound tracing. The mean value of the three trials was calculated and taken to be the wound surface area.
Change in wound volume | Baseline and six weeks after the intervention
  Assessment of wound volume was done by saline injection tool. A syringe of twenty cubic centimeters filled with normal sterilized saline was used. The patient was positioned in a comfortable position that allows the wound to be filled with the saline solution maximally. The saline was injected into each wound until its filling. The amount of saline injected was detected in cubic centimeters. These measurements were conducted for each patient before and after of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Shaimaa MA Elsayeh, PhD, Study Director — Lecturer at Faculty of Physical Therapy, Cairo University
Locations (1):
- Shaimaa Mohamed Ahmed Elsayeh, Cairo, New Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No